CLINICAL TRIAL: NCT02606292
Title: Photoacoustic Endoscopy of Barrett's Esophagus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201204145
Record Dates: First submitted 2015-11-09; First posted 2015-11-17 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Standard of Care; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: PAE assessment (Experimental): -The PAE-EUS assessment will be performed in the operating room by the after induction of general anesthesia and following strict sterile technique while the patient is being positioned and prepped for esophageal surgery.
  Interventions: Procedure: Photoacoustic endoscopy; Procedure: Endoscopic ultrasound (standard of care); Procedure: Endoscopic surgery (standard of care)

INTERVENTIONS:
Procedure: Photoacoustic endoscopy
  Other Names: PAE
Procedure: Endoscopic ultrasound (standard of care)
  Other Names: EUS
Procedure: Endoscopic surgery (standard of care)

SUMMARY:
Endoscopy is an important technique in medicine to diagnose internal organs. Video endoscopy has been the most common technique providing clear, real time video images of organs' surfaces. However, this technique only images the surface and cannot effectively diagnose diseased tissues that develop in endothelial tissues. Endoscopic ultrasound (EUS) has been developed to overcome this limitation, and it is widely utilized in diagnosing GI diseases. This technique can image very deep areas of organs, up to several centimeters; however, it suffers from speckle artifacts and cannot adequately provide early diagnosis of tissue abnormalities that do not show mechanical properties that differ significantly from those of normal tissues.

The investigators propose that photoacoustic endoscopy (PAE), an endoscopic embodiment of the rapidly growing photoacoustic tomography (PAT) technology, can fulfill the aforementioned need.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older.
* Patients with Barrett's esophagus scheduled for esophageal surgery.
* Patients with GERD, but without Barrett's esophagus, scheduled for esophageal surgery.
* Subjects must be able to understand and willing to sign a written informed consent form.

Exclusion Criteria:

* Inability to give informed consent.
* Pregnancy.
* Age less than 18 years
* Previous esophageal procedure (surgery, photodynamic therapy, argon plasma coagulation, endoscopic mucosal resection).
* Acute GI bleeding.
* Coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of PA endoscopic imaging as an alternative real-time noninvasive tool for evaluation of Barrett's esophagus as measured by the agreement between the PA imaging system and the standard esophageal biopsy for diagnosing Barrett's epithelium | Day 1
  -The investigators will image a series of human esophagi in patients with an established diagnosis of Barrett's esophagus with/without dysplasia to fine-tune the PA imaging system. The investigators will assess the agreement between the PA imaging system and the standard clinical practice of four-quadrant esophageal biopsy previously performed in this cohort of patients as part of his/her active surveillance program.
Sensitivity and specificity of PA endoscopic imaging for identification of Barrett's epithelium compared to esophageal biopsy | Day 1
  -The investigators will image a series of human esophagi in patients with an established diagnosis of Barrett's esophagus with/without dysplasia to fine-tune the PA imaging system. The investigators will assess the agreement between the PA imaging system and the standard clinical practice of four-quadrant esophageal biopsy previously performed in this cohort of patients as part of his/her active surveillance program.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan F Meyers, M.D., M.P.H., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu